CLINICAL TRIAL: NCT07039591
Title: A Randomized Open Label Crossover Trial to Assess Performance Attributes and Acceptability of Non-medicated Intravaginal Rings Among Sexually Active Women in Atlanta, GA
Brief Title: Assess Performance Attributes and Acceptability of Non-medicated Intravaginal Rings Among Sexually Active Women in Atlanta, GA
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CBR-001
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proto-type IVR (Experimental): 60 women comparing acceptability of three different non-medicated IVRs (2 silicone and 1 EVA) based on the Intravaginal Ring Acceptability Scale (IVR-AS).
  Interventions: Device: Pro-type IVR

INTERVENTIONS:
Device: Pro-type IVR — Women will test three non-medicated IVRs on two one-day clinic visits (two on the first day, one on the second day) by manipulating them, vaginally inserting each ring and then performing a controlled set of tasks simulating routine daily activities with the ring in the vagina.

SUMMARY:
A randomized open label crossover trial to assess performance attributes and acceptability of non-medicated intravaginal rings among sexually active women in Atlanta, GA

ELIGIBILITY:
Inclusion Criteria:

* 1. Cisgender female aged 18-49 years old, inclusive, at screening based on self-report.

  2. Sexually active, defined as having penile-vaginal sex at least once a week, on average, over the past three months with the same male partner, and intends to continue having sexual intercourse at the current frequency for at least three months.

  3. Healthy based on medical history, physical exam (including pelvic exam with visual inspection) at screening.

  4. Using effective non-vaginal method of contraception (oral contraception, injectable, patch, IUD, sterilization, male condoms) 5. Competent to provide written informed consent based on Investigator's assessment.

  6. Agrees to not participate in any other clinical research involving investigational or marketed products for the duration of this trial.

Exclusion Criteria:

* 1. Known or suspected allergy to silicone or EVA, as reported by participant. 2. Positive pregnancy test at screening or enrollment based on urine hCG test. 3. Positive for HIV at screening based on rapid test per site SOPs. 4. Presence of any clinically significant genital epithelial findings (e.g. abrasions, ulcerations, lacerations, or vesicles) at screening.

  5. Positive chlamydia, gonorrhea, or trichomoniasis test at screening. 6. Symptomatic vulvovaginal candidiasis, bacterial vaginosis (BV), or urinary tract infection (UTI) at screening. (Participants who are symptomatic at initial screening will be referred for testing and treatment and may be reconsidered for eligibility after completing treatment and/or if no longer symptomatic).

  7. Presence of genital abnormalities on visual exam with speculum that would contraindicate IVR use.

  8. History of significant uterine or vaginal prolapse, or urethral obstruction. 9. Unexplained vaginal bleeding per self-report within the last three months. 10. Currently breastfeeding per self-report. 11. Partial or complete hysterectomy per self-report. 12. History of gynecological surgery in the six months prior to screening per self-report.

  13. Within six weeks post abortion or six months postpartum, per self-report. 14. Using vaginal contraception (diaphragm, female condom, spermicide, IVR). 15. Known current drug abuse, including illicit drugs, or alcohol abuse. 16. Any other condition the clinician feels would jeopardize the health and wellbeing of the participant after assessing the participant's potential eligibility for the study.

  17. Unable to comply with study requirements, including but not limited to, attending all study visits and using the IVRs as directed.

  18. Participation in any other clinical research trial involving investigational or marketed products currently or within one month of participation prior to screening, including any trial of a spermicide, microbicide and/or drug.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Mean Acceptability Score per IVR | From enrollment to the end of treatment at approximately 13 weeks
  For the primary outcome we will compute the mean acceptability score per IVR, for each of three IVRs of different compression strengths. The scores women give each of the three rings will be compared using a mixed-effects model with orthogonal contrasts, with all 3 pairwise comparisons using the Bonferroni method to adjust for multiple comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided